CLINICAL TRIAL: NCT03134300
Title: Cytokine Persistence as a Marker of Inflammation in the at Risk, Low Socioeconomic Status Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Arvind Chandrakantan, Assistant Professor of Anesthesiology & Pediatrics, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-39874
Record Dates: First submitted 2017-04-19; First posted 2017-04-28 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Obstructive Sleep Apnea of Child

STUDY DESIGN:
Intervention Model Description: 2 groups for the same intervention (AT), one from low SES, one from high SES. Cytokine draw periprocedurally, and 3 weeks post procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low SES (Active Comparator)
  Interventions: Diagnostic Test: Cytokine from blood
- Normal/high SES (Placebo Comparator)
  Interventions: Diagnostic Test: Cytokine from blood

INTERVENTIONS:
Diagnostic Test: Cytokine from blood — Blood draw- one intraoperative, one 3 weeks postoperative

SUMMARY:
The investigators wish to study the role of persistent markers of inflammation in executive function in young children during critical periods of synaptogenesis (ages 2-3). While the role of markers of inflammation have been validated in the pathogenesis in multiple disorders in the adult population, their study in pediatrics is limited. The investigators therefore propose that demonstration of persistent cytokine inflammatory markers in this preliminary study will allow larger studies to proceed.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common multisystem disorder, affecting up to 10% of the pediatric population. There is scant data about OSA and adenotonsillectomy (AT) outcomes in the very young (ages 1-3). Young children with moderate/severe OSA are often underprivileged, low socioeconomic status (SES) minorities with limited access to care. Further complicating the problem is that African American children may suffer a higher preoperative and post-AT burden of disease, with greater negative consequences to these vulnerable children. Up to 75% of children with OSA continue to have sequelae of the disease post-AT. These include poor school performance, delayed speech, inattention, and long term neurocognitive dysfunction. It has been demonstrated that younger patients (below the age of 3) have larger tonsils and stunted growth on presentation for AT. More telling is that younger children face greater morbidity from the procedure, including respiratory complications, postoperative bleeding, and perioperative anoxic/hypoxic injury as validated by multiple studies. A recent study studied watchful waiting versus early AT in two groups of patients aged 5-9 without severe OSA. The findings indicated that early AT improved respiratory and quality of life indices without corresponding improvement in attention or cognitive function as assessed by neuropsychological testing 7 months post intervention. So it leads to the further question of whether children with severe OSA truly benefit from the procedure at all, and whether there maybe a trend towards harm. In this particular scenario, the investigators are hypothesizing that serum based biomarkers in the form of cytokines are of significant diagnostic benefit in demonstrating ongoing inflammation.

Therefore, the surgical stimulus and consequent stress response in the form of centrally mediated cytokines and inflammatory mediators demands study. These has been well analyzed with adult acute and chronic pain, and have been associated with neurocognitive impairment, but have not been studied as a neurocognitive biomarker in the pediatric population. Children from lower SES, with less stable social environments, or other cultural/linguistic barriers are higher risk and urgently require study.

ELIGIBILITY:
Inclusion Criteria: OSA for adenotonsillectomy -

Exclusion Criteria:

-

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Increased cytokines in low SES group | 3 weeks post operative

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Chandrakantan, MD, MBA, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No